CLINICAL TRIAL: NCT06307041
Title: Effects of 0.2% Hyaluronic Acid Gel-Impregnated Dental Flosses on Clinical Gingival Parameters: A Randomized Clinical Trial
Brief Title: Effects of 0.2% Hyaluronic Acid Gel-Impregnated Dental Flosses on Clinical Gingival Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem SARAÇ ATAGÜN (Other)
Responsible Party: Sponsor-Investigator, Özlem SARAÇ ATAGÜN, assistant professor, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSATAGUN
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Gingivitis
Keywords: Hyaluronic Acid; Dental Floss; Gingivitis; Oral Hygiene
MeSH Terms: conditions — Gingivitis | interventions — Dental Devices, Home Care

STUDY DESIGN:
Intervention Model Description: single-center, single-blinded, split-mouth, randomized clinical trial
Who Masked: Investigator
Masking Description: The investigator who performed the measurements was blinded to which side of patients was the test group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (HA group) (Other): One side is HA gel impregnated dental floss usage
  Interventions: Device: Dental floss+Gengigel
- Control Group (Other): One side is dental floss usage
  Interventions: Device: Dental Floss

INTERVENTIONS:
Device: Dental floss+Gengigel — 0.2% Hyaluronic Acid Gel-Impregnated Dental Flosses
  Arms: Test (HA group)
Device: Dental Floss — Dental Flosses
  Arms: Control Group

SUMMARY:
This study aimed to evaluate the effects of 0.2% HA-impregnated dental flosses on the clinical periodontal parameters of patients with gingivitis.

DETAILED DESCRIPTION:
Gingivitis is a common inflammatory lesion caused by the build-up of oral biofilm and is an essential precursor to periodontitis. For its treatment, oral hygiene habits, such as dental flossing, must be improved, and adjunctive materials, such as hyaluronic acid, may be used to reduce plaque formation and gingival inflammation. This study aimed to assess the effects of 0.2% hyaluronic acid gel (Gengigel®)-impregnated dental flosses on the clinical periodontal markers of patients with gingivitis.

This clinical study adopted a split-mouth, randomized controlled trial design. After clinical data were assessed at baseline, and supragingival scaling and planing was performed, bilateral gingivitis regions were randomly allocated to either a test group (hyaluronic acid gel-impregnated floss) or a control group (regular floss) using a computer-generated randomization table. Clinical parameters were recorded at 1, 2, and 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18-55 years of age
2. Being systemically healthy
3. Having gingivitis
4. Not to have used any medication in the last three months
5. Not smoking
6. Right-handed
7. At least 20 natural teeth

Exclusion Criteria:

1. Patients with interdental caries
2. Patients with orthodontic appliances
3. Patients with removable (partial) prostheses
4. Patients with oral and/or peri-oral pain
5. Patients with significant oral lesions
6. Patients with antibiotic use in the last 3 months, pregnancy and breastfeeding
7. Patients who have undergone periodontal treatment within the last 6 months

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Clinical Periodontal Parameter-Gingival Index (GI) | Baseline-4 weeks
  Improvement in GI (lower scores mean a better outcome)Minimum score:0 Max.score:3
Clinical Periodontal Parameter-Papillary Bleeding Index (PBI) | Baseline-4 weeks
  Improvement in PBI (lower scores mean a better outcome)Minimum score:0 Max.score:4
Clinical Periodontal Parameter-Plaque Index(PI) | Baseline-4 weeks
  Improvement in PI (lower scores mean a better outcome)Minimum score:0 Max.score:5

CONTACTS AND LOCATIONS:
Overall Officials: özlem saraç atagün, PhD, Principal Investigator — Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi Periodontoloji AD
Locations (1):
- Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atagun OS, Sen SC, Ustaoglu G, Ozcan E. Effects of 0.2% Hyaluronic Acid Gel-Impregnated Dental Floss on Clinical Gingival Parameters: A Randomised Clinical Trial. Int J Dent Hyg. 2025 May;23(2):312-318. doi: 10.1111/idh.12856. Epub 2024 Oct 29. PMID 39473003